CLINICAL TRIAL: NCT02246283
Title: Schizophrenia for "Life" - a Registry and Interview Study Among Elderly With Lifelong Schizophrenia
Status: Completed | Type: Observational
Sponsor: Kjeld Andersen (Other)
Collaborators: The Psychiatric Research Foundation in Southern Denmark (Unknown); Region of Southern Denmark (Other); University of Southern Denmark (Other); The Danish Mental Health Foundation (Other); The Danish Health Foundation (Helsefonden) (Unknown); The non-profit foundation Trygfonden. (Unknown); Odense Patient Data Explorative Network (Other); Jeppe Juhl and Ovita Juhls Memorial Grant (Unknown); Butcher Max Wørzner and wife Inger Wørzner's Memorial Grant (Unknown)
Responsible Party: Sponsor-Investigator, Kjeld Andersen, Professor, University of Southern Denmark
Organization: University of Southern Denmark (Other)
Other Study IDs: Schizophrenia-Lifelong
Record Dates: First submitted 2014-09-17; First posted 2014-09-22 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Schizophrenia
Keywords: schizophrenia; elderly; lifelong; quality of life; register; questionaire
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The elderly demographic is on the rise - and this includes elderly living with schizophrenia. Yet very little is known about their lives, how they cope with their condition and how it develops over time.

Research in this patient-group is sparse; overall there seem to be a tendency for elderly patients to manifest fewer psychotic symptoms and experiencing an increase in the psychological quality of life with older age. Opinions are divided on the degree and extent to which this tendency reflects remission and/or recovery in older patients.

In order to identify factors associated with a positive outcome we:

* Investigate the course and the outcomes of the illness over the lifespan, as well as the life course and outcomes.
* Investigate the current status of mental and physical health, quality of life as well as functional competence of elderly (55+ yr) with schizophrenia.

Also the investigators

- Compare the trajectory and prognosis of schizophrenia (a chronic mental illness) with type 1 diabetes (a chronic somatic illness).

This study will yield vital insights into how schizophrenia develops over time, isolating factors that determine how well patients fare. The perspective is to advance knowledge of elderly with schizophrenia with a view to optimizing and increasing the effectiveness of the interventions offered to this group.

ELIGIBILITY:
Inclusion Criteria:

Initial schizophrenia diagnosis between the ages 18-40 (both incl) in the period 1970-1979 (both incl) Interview study: Residence in Region of Southern Denmark

Exclusion Criteria:

Interview study: Mental retardation

-

Ages: 55 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Registry study: A nationwide register cohort study (1970-79) identifying psychiatric admissions (aged 18-40), who were registered with a schizophrenia diagnosis. Several Danish registers are applied.
  Interview study: A cross-sectional survey where 150 randomly drawn surviving members of the register cohort resident in the Region of Southern Denmark will be interviewed on the basis of internationally validated assessment tools.
Sampling Method: Non-Probability Sample
Enrollment: 10404 (Actual)
Dates: Start 2013-09; Primary Completion 2015-09 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Ageing with schizophrenia | up to 45 years
  Prognosis measured by use of healthcare system, use of medicine, co-morbidity, mortality, causes of mortality, and socio-demographic data, including highest level of education, years of employment/un-employment, use of health- and welfare services.

SECONDARY OUTCOMES:
Quality of life | 1 month
  Questionnaire
Remission | 6 months
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Maria Brink, MD, Principal Investigator — University of Southern Denmark
Locations (1):
- Research Unit of Psychiatry, Psychiatric Unit Odense - University function, Odense C, Denmark